CLINICAL TRIAL: NCT00047710
Title: A Phase I Trial of Concurrent RHUMAB VEGF (BEVACIZUMAB) and Capecitabine-based Chemoradiation for Patients With Locally Advanced Pancreatic Cancer
Brief Title: Study of Combined RHUMAB VEGF and Capecitabine-based Chemoradiation for Patients With Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-146
Record Dates: First submitted 2002-10-14; First posted 2002-10-16 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; pancreas cancer; pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bevacizumab; Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab (Experimental): Radiation, Bevacizumab, and Capecitabine
  Interventions: Drug: Bevacizumab; Drug: Capecitabine; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Bevacizumab — Beginning 2 weeks prior to radiotherapy, dose of 5 mg/kg by vein then of 2.5 mg/kg during radiotherapy for four weeks every 2 weeks (three doses).
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Capecitabine — 650mg/m^2 taken by mouth twice a day 15-52 during the radiotherapy.
  Other Names: Xeloda
Radiation: Radiotherapy — Radiography given once a day for 5 days at 50.4 Gy in 28 fractions over 5.5 weeks.
  Other Names: XRT

SUMMARY:
The goal of this clinical research study is to find the highest safe dose of the drug Bevacizumab that can be given in combination with chemoradiation for the treatment of pancreatic cancer. The effect that this combination treatment has on the tumor will also be studied.

DETAILED DESCRIPTION:
This study administers 50.4 Gy of radiation for unresectable pancreatic cancer with concurrent capecitabine and an experimental drug, Bevacizumab. The drug is an antiangiogenic agent (kills tumor blood vessels) and has been shown in preclinical models to enhance the antitumor effect of radiation and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Cytology or histologic proof of adenocarcinoma of the pancreatic head, body or tail prior to treatment.
* Patients with nonmetastatic, unresectable, disease are eligible.
* Patients with regional nodal disease are eligible.
* Karnofsky performance status >/=70.
* No upper age restriction.
* Absolute granulocyte count >1,500 cells/mm3 and platelet count at least 100,000 cells/mm3.
* Serum bilirubin less than 5mg/dl prior to the start of therapy with adequate biliary decompression.
* Adequate bilateral renal function.
* Serum creatinine <1.5 mg/dl.
* Adequate liver function; Alanine aminotransferase (ALT)/aspartate aminotransferase (AST)</=5 times upper limit of normal.
* Sexually active men must practice contraception during study.
* Patients must sign study-specific consent form.

Exclusion Criteria:

* History or evidence upon physical examination of CNS disease.
* Active infection requiring parenteral antibiotics on Day 0. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study.
* Current or recent use of full-dose oral or parenteral anticoagulants or thrombolytic agent.
* Chronic, daily treatment with aspirin or nonsteroidal anti-inflammatory medications.
* Pregnancy or lactation.
* Proteinuria at baseline or impairment of renal function.
* Serious, nonhealing wound, ulcer, or bone fracture.
* Evidence of bleeding diathesis or coagulopathy
* Clinically significant cardiovascular disease, congestive heart failure, serous cardiac arrhythmia requiring medication, or significant peripheral vascular disease within 1 year prior to Day 0.
* History of aneurysms, strokes, transient ischemic attacks, and arteriovenous malformations.
* Serous concomitant medical or psychiatric disorders.
* Cohort receiving Capecitabine

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2002-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Safety of combination Radiation, Bevacizumab, and Capecitabine. | 6 weeks after the completion of therapy

SECONDARY OUTCOMES:
To evaluate the local tumor response and median survival in patients treated with the above regimen. | 6 weeks after the completion of therapy.
To evaluate VEGF serum levels before and after anti-VEGF therapy. | 6 weeks after the completion of therapy.
To evaluate tumor hypoxia via PET scanning (gallium PET with the novel hypoxia tracer Ga-68 ECMN) before, during, and after therapy. | 6 weeks after the completion of therapy.
To evaluate quality of life in patients receiving this therapy. | 6 weeks after the completion of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher H. Crane, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MDAnderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org